CLINICAL TRIAL: NCT01790659
Title: A Randomized, Double-blind, Pivotal Phase 3 Study of WR 279,396 (Paromomycin + Gentamicin Topical Cream) and Paromomycin Alone Topical Cream for the Treatment of Cutaneous Leishmaniasis in Panama
Brief Title: Phase 3 Study of Walter Reed (WR) 279,396 and Paromomycin Alone for the Treatment of Cutaneous Leishmaniasis in Panama
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-12-21
Record Dates: First submitted 2013-02-05; First posted 2013-02-13 (Estimated); Results first posted 2017-08-23 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Cutaneous Leishmaniasis
Keywords: leishmaniasis; cutaneous leishmaniasis; Leishmania panamensis; L panamensis; Paromomycin; Paromomycin/Gentamicin
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Paromomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WR 279,396 (Experimental): (Paromomycin and Gentamicin Topical Cream)
  Interventions: Drug: WR 279,396
- Paromomycin (Experimental): Paromomycin alone
  Interventions: Drug: Paromomycin

INTERVENTIONS:
Drug: WR 279,396 — WR 279,396 is a topical cream of paromomycin 15% and gentamicin 0.5%
  Other Names: Paromomycin/Gentamicin topical cream
  Arms: WR 279,396
Drug: Paromomycin — Paromomycin alone
  Arms: Paromomycin

SUMMARY:
This study is a pivotal Phase 3, randomized, double-blind, 3-site, two-group trial assessing the efficacy and safety of WR 279,396 Topical Cream and Paromomycin Alone Topical Cream in subjects with CL in Panama. The primary objective of this study is to determine if WR 279,396 results in statistically superior final clinical cure rates of an index lesion when compared with Paromomycin Alone for the treatment of CL in Panama expected to be caused by L panamensis.

DETAILED DESCRIPTION:
Subjects will be recruited from three regions in Panama known to be endemic for L panamensis CL. Subjects will be screened over a period up to 28 days for eligibility including medical history, physical examination, leishmaniasis history, vital signs, clinical chemistry, prior medications, and parasitology for confirmation of ulcerative CL. If eligible, subjects will be randomized in a targeted 1:1 ratio (200 subjects per group) using site as a stratification variable to receive either WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) or Paromomycin Alone (15% paromomycin topical cream) by topical application to CL lesions once daily for 20 days. Efficacy will be assessed by measuring the size of the index lesion ulcer, non-index lesions ulcers, and overall size of other non-ulcerated lesions at baseline (before the start of treatment), and on Study Days 20, 35 ± 2 days, 49 ± 4 days, 63 ± 7 days, 100 ± 14 days, and 168 ± 14 days. A notation will be made if clinical evidence of parasite persistence is observed at the Day 63 and beyond visits including significant erythema and induration when a lesion has otherwise completely re-epithelialized to document any subjects removed from the study early if the investigator judges them to be in need of rescue treatment. A photograph will be taken of all lesions at baseline, Day 20 and each of the follow-up visits. Safety will be assessed by monitoring adverse events (AEs) from the start of treatment until study completion, lesion site reactions during treatment, physical examination of the nasal and oral mucosa for appearance of mucosal leishmaniasis on Days 63 ± 7 days, 100 ± 14 days, and 168 ± 14 days, concomitant medication use for the duration of the study, blood creatinine, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels on Study Day 20. After the sponsor's approval, biochemistry can be repeated in the case of abnormal results and if the causes of these results could not be determined. A repeat pregnancy test on Day 35. Recent infection with leishmaniasis prior to the start of the study may result in the development of lesions that were not present at the start of the study that did not receive treatment. New lesions may be treated at the discretion of the investigator with the topical cream to which the subject was assigned any time during the conduct of the study except that treatment must be completed by the Day 168 visit. If a new lesion is discovered at the final study visit, the subject will be referred to their primary physician for treatment.

Subjects who fail therapy (see definition of failure below) will be taken off study and may be administered rescue therapy at the discretion of the subject's personal physician. If the subject met the criteria for therapy failure but was undergoing treatment for new lesions, the subject can continue in the study (by signing a consent addendum) if the investigator decides it is in the best interest of the subject to do so.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 2 years-of-age
* Subject or legal guardian able to give written informed consent or assent, as appropriate
* Diagnosis of CL in at least one lesion by at least one of the following methods: 1) positive culture for promastigotes or 2) microscopic identification of amastigotes in stained lesion tissue
* At least one ulcerative lesion ≥ 1 cm and ≤ 5 cm that has a diagnosis of CL
* Willing to forego other forms of treatments for CL including other investigational treatments during the study
* In the opinion of the investigator, subject (or their legal guardian), subject is capable of understanding and complying with the protocol
* If female and of child-bearing potential, must have a negative serum pregnancy test during screening and agree to use an acceptable method of birth control during the treatment phase and for 1 week after treatment is completed

Exclusion Criteria:

* Lesion due to leishmania that involves the nasal or oral mucosa or any signs of mucosal disease that might be due to Leishmania
* Only a single lesion on the ear with erosive cartilage
* Signs and symptoms of disseminated disease in the opinion of the investigator
* More than 10 lesions
* Female who is breast-feeding
* Significant organ abnormality, chronic disease such as diabetes, severe hearing loss, evidence of renal or hepatic dysfunction, or creatinine, aspartate aminotransferase (AST), or alanine aminotransferase (ALT) greater than 15% above the upper limit of normal (ULN) as defined by the clinical laboratory defined normal ranges
* Received treatment for leishmaniasis including any medication with pentavalent antimony including sodium stibogluconate (Pentostam™), meglumine antimoniate (Glucantime™); amphotericin B (including liposomal amphotericin B and amphotericin B deoxycholate); or other medications containing paromomycin (administered parenterally or topically) or methylbenzethonium chloride (MBCL); gentamicin; fluconazole; ketoconazole; pentamidine; miltefosine, azithromycin or allopurinol that was completed within 56 days of starting study treatments
* History of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Sosa, MD, FACP, Principal Investigator — Instituto Conmemorativo Gorgas de Estudios de la Salud
Locations (1):
- Instituto Conmemorativo Gorgas de Estudios de la Salud,, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from three regions in Panama. Subjects were screened over a 28 day period.
Period: Overall Study
Arm/Group | WR 279,396 | Paromomycin
Started | 201 | 198
Completed | 195 | 192
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WR 279,396 | Paromomycin | Total
Number analyzed (Participants) | 201 | 198 | 399
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96 | 88 | 184
  Between 18 and 65 years | 105 | 110 | 215
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (16.8) | 23.6 (15.1) | 23.2 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 149
  Male | 125 | 125 | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 201 | 196 | 397
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 198 | 192 | 390
  Unknown or Not Reported | 3 | 6 | 9
Number of baseline lesions [Mean (Standard Deviation); unit: Lesions] | 2.27 (1.71) | 2.13 (1.63) | 2.20 (1.67)
Lesion sizes [Mean (Standard Deviation); unit: mm] — Lesion size was calculated in mm
  mm | 120 (146) | 121 (152) | 120 (149)
Length of time between initial presence current lesions and treatment [Mean (Standard Deviation); unit: Days] — Length of time in days before treatment that lesions were first noticed
  Days | 59.7 (53.6) | 62.1 (57.7) | 60.9 (55.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Final Clinical Cure
Description: The primary efficacy endpoint is percent of subjects with final clinical cure. Final clinical cure is defined as follows:
  * Subject has initial clinical cure (100% re-epithelialization of index lesion by nominal Day 63); OR,
  * Subject has initial clinical improvement (> 50% re-epithelialization of index lesion by nominal Day 63) followed by 100% re-epithelialization of the index lesion on or before nominal Day 100; AND,
  * Subject has no relapse of index lesion.
Time Frame: baseline (before the start of treatment), and on Study Days 20, 35 ± 2 days, 49 ± 4 days, 63 ± 7 days, 100 ± 14 days, and 168 ± 14 days
Population: MITT subjects
Measure: Number; unit: percent of participants
Arm/Group | WR 279,396 | Paromomycin
Number analyzed (Participants) | 201 | 198
percent of participants | 78.6 | 77.8

2. Secondary Outcome: Percentage of Subjects With All Lesions Cured
Description: • Percentage of subjects with all lesions cured, defined as: Final clinical cure as defined in primary objective (which is based solely on the index lesion); AND, Cure of all other lesions by nominal Day 100 (100% re-epithelialization of all ulcerated lesions and resolution of all other types of lesions)
Time Frame: 100 ± 14 days
Population: MITT subjects
Measure: Number; unit: percentage of participants
Arm/Group | WR 279,396 | Paromomycin
Number analyzed (Participants) | 201 | 198
percentage of participants | 75.1 | 76.3

3. Secondary Outcome: Percentage of All Lesions Cured at Day 168 (Ignores Per Subject Cure Rate)
Description: Percentage of all lesions meeting criteria for clinical cure during the study at 168 day mark for mITT subjects
Time Frame: Day 168
Population: Cure rates of all lesions over time without regard to subject for mITT subjects
Measure: Number; unit: percentage of lesions
Arm/Group | WR 279,396 | Paromomycin
Number analyzed (Participants) | 201 | 198
percentage of lesions | 77.2 | 83.3

4. Secondary Outcome: Area of Ulceration (mm^2) of the Index Lesion at Each Measurement Time Point
Description: Area of ulceration (mm^2) of the index lesion at each measurement time point for mITT subjects
Time Frame: as for outcome 1
Population: mITT subjects
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | WR 279,396 | Paromomycin
Number analyzed (Participants) | 201 | 198
mm^2
  Day 1 | 153 (137) | 165 (167)
  Day 20 | 831 (627) | 928 (986)
  Change from baseline Day 20 | 677 (602) | 762 (933)
  Day 35 | 68.3 (138) | 96.1 (188)
  Change from baseline Day 35 | -84.1 (156) | -69.9 (172)
  Day 49 | 29.4 (87.2) | 33.9 (100)
  Change from baseline Day 49 | -123 (144) | -132 (157)
  Day 63 | 29.9 (119) | 27.6 (107)
  Change from baseline Day 63 | -123 (167) | -136 (171)
  Day 100 | 12.5 (85.9) | 7.41 (56.9)
  Change from baseline Day 100 | -144 (163) | -152 (165)
  Day 168 | 13.3 (111) | 1.37 (9.89)
  Change from baseline Day 168 | -147 (171) | -160 (161)

5. Secondary Outcome: Area of Ulceration (mm^2) All Treated Lesions at Each Measurement Time Point
Description: Area of ulceration (mm^2) of all treated lesions from baseline (before the start of treatment), and on Study Days 20, 35 ± 2 days, 49 ± 4 days, 63 ± 7 days, 100 ± 14 days, and 168 ± 14 days for mITT subjects. Data presented is as presented in the Final Clinical Study Report; any inconsistencies can't be changed.
Time Frame: as for outcome 1
Population: All lesions for mITT Subjects
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Number of lesions
Arm/Group | WR 279,396 | Paromomycin
Number analyzed (Participants) | 201 | 198
Number analyzed (Number of lesions) | 457 | 422
mm^2
  Day 1 | 115 (152) | 115 (149)
  Day 20 | 656 (683) | 699 (897)
  Change from baseline Day 20 | 533 (632) | 577 (829)
  Day 35 | 53.0 (132) | 66.1 (159)
  Change from baseline Day 35 | -62.8 (167) | -51.9 (146)
  Day 49 | 21.4 (76.8) | 23.9 (88.2)
  Change from baseline Day 49 | -93.8 (160) | -92.1 (132)
  Day 63 | 19.9 (94.6) | 15.8 (82.3)
  Change from baseline Day 63 | -96.2 (170) | -98.7 (142)
  Day 100 | 7.49 (58.8) | 4.64 (42.8)
  Change from baseline Day 100 | -113 (166) | -109 (143)
  Day 168 | 9.14 (87.7) | 0.83 (7.23)
  Change from baseline Day 168 | -118 (182) | -114 (147)

6. Secondary Outcome: Median Time to Initial Clinical Cure for Index Lesions
Description: Median time to initial clinical cure for index lesions (100% re-epithelialization of the index lesion)
Time Frame: When 100% re-epithelialization of the index lesion is observed at any visit Study Days (20, 35 ± 2 days, 49 ± 4 days, 63 ± 7 days, 100 ± 14 days, and 168 ± 14 days
Population: MITT subjects
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | WR 279,396 | Paromomycin
Number analyzed (Participants) | 201 | 198
Days | 36.000 [35 to 49] | 48.000 [36 to 49]

ADVERSE EVENTS:
Time Frame: AE's were assessed at baseline, days 2-9 daily, day 20, 35, 49, 63, 100, and 168 (applicable)
Description: AE's including application site reactions including elicited examination for pain, and clinician examination for erythema/redness, swelling/edema and vesicles. Physical examination findings of evidence of mucosal leishmaniasis will be reported as an AE.
Arm/Group | WR 279,396 | Paromomycin
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/198
Serious Adverse Events (participants affected / at risk) | 2/201 | 1/198
Other Adverse Events (participants affected / at risk) | 201/201 | 198/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WR 279,396 (N=201) | Paromomycin (N=198)
Second degree burn: scalding water (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Infection of surgical site (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WR 279,396 (N=201) | Paromomycin (N=198)
Lymphadenitis (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 10 (10)
Abdominal pain (upper) (Gastrointestinal disorders) | 5 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 4 (4)
Gastritis (Gastrointestinal disorders) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Application site dermatitis (General disorders) | 21 (21) | 13 (13)
Application site erosion (General disorders) | 4 (4) | 7 (7)
Application site erythema (General disorders) | 2 (2) | 3 (3)
Application site injury (General disorders) | 22 (22) | 38 (38)
Application site pain (General disorders) | 14 (14) | 16 (16)
Application site pruritus (General disorders) | 11 (11) | 8 (8)
Mucosal erosion (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Conjunctivitis (Infections and infestations) | 2 (2) | 4 (4)
Cutaneous Leishmaniasis (Infections and infestations) | 10 (10) | 12 (12)
Folliculitis (Infections and infestations) | 9 (9) | 14 (14)
Gastroenteritis (Infections and infestations) | 10 (10) | 9 (9)
Lymphangitis (Infections and infestations) | 29 (29) | 16 (16)
Mucocutaneous Leishmaniasis (Infections and infestations) | 5 (5) | 7 (7)
Nasopharyngitis (Infections and infestations) | 126 (126) | 112 (112)
Pharyngitis (Infections and infestations) | 9 (9) | 8 (8)
Pyoderma (Infections and infestations) | 3 (3) | 4 (4)
Rhinitis (Infections and infestations) | 12 (12) | 13 (13)
Superinfection bacterial (Infections and infestations) | 20 (20) | 19 (19)
Arthrpod bite (Injury, poisoning and procedural complications) | 21 (21) | 15 (15)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Limb Injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 37 (37) | 22 (22)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 99 (99) | 97 (97)
Pruritus (Skin and subcutaneous tissue disorders) | 60 (60) | 53 (53)
Skin erosion (Skin and subcutaneous tissue disorders) | 25 (25) | 13 (13)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No